CLINICAL TRIAL: NCT04279392
Title: Feasibility of Bisphosphonate Use on Sleeve Gastrectomy Associated Bone Loss: Healthy Body, Healthy Bones Trial
Brief Title: Healthy Body, Healthy Bones After Bariatric Surgery Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0820-19-FB
Record Dates: First submitted 2020-01-31; First posted 2020-02-21 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Bariatric Surgery Candidate; Bone Loss; Bone Resorption
MeSH Terms: conditions — Bone Diseases, Metabolic; Bone Resorption | interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial each subject will be randomized (1:1, block randomization with a block size of 10) to one treatment group (Active or Inactive treatment) and will be considered part of the intent-to-treat (ITT) cohort. The research pharmacist will be responsible for completing the randomization process, and will hold the group assignment data. All other study personnel will be blinded to group assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research pharmacist will deliver the drug pr placebo to the treatment nurse in an unlabeled 100 ml saline bag for infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Infusion (Active Comparator): At 6 weeks post surgery, 5 mg of zoledronic acid in 100 ml of saline will be infused intravenously over a 15 minute time period.
  Interventions: Drug: Zoledronic Acid 5 mg/Bag 100 ml Inj
- Non-active Infusion (Placebo Comparator): At 6 weeks post surgery, 100 ml of saline will be infused intravenously over a 15 minute time period.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Zoledronic Acid 5 mg/Bag 100 ml Inj — Zoledronic acid infusion
  Other Names: Reclast
  Arms: Active Infusion
Drug: Placebos — Saline infusion
  Arms: Non-active Infusion

SUMMARY:
One in three adults in the United States suffers from obesity. Bariatric surgery is an increasingly utilized and effective treatment for obesity and obesity-related comorbidities, however, the massive weight loss associated with bariatric surgery adversely affects bone leads to an increased risk of fracture. Bisphosphonate medications, such as zoledronic acid, are used to treat bone loss in patients with osteoporosis, and this study investigates whether this medication can prevent bone loss associated with surgical weight loss procedures.

DETAILED DESCRIPTION:
One in three adults in the United States suffers from obesity. Bariatric surgery is an increasingly utilized and effective treatment for obesity and obesity-related comorbidities, however, the massive weight loss associated with bariatric surgery adversely affects bone metabolism. Significant decreases in bone mineral density lead to an increased risk of fracture and subsequent reduction in physical function among bariatric surgery patients. Bisphosphonate medications, such as zoledronic acid, have been evaluated for safety and efficacy in combating bone loss in patients with osteoporosis, but their use in bariatric surgery-induced bone loss has not been explored. The primary goal of this study is to investigate whether bisphosphonate therapies are able to combat bone loss associated with surgical weight loss procedures. This research proposal is a 1-year, pilot randomized controlled trial (RCT) involving 30 adult sleeve gastrectomy patients randomized to receive either a one-time zoledronic acid infusion or placebo (n=15 per group). The investigators hypothesize that zoledronic acid, a standard treatment for low bone density, will be an effective intervention to reduce sleeve gastrectomy-induced bone loss. Bone loss is an unintended consequence of an otherwise life-saving procedure, with declining bone health potentially contributing to major morbidity in those undergoing a bariatric procedure. Identifying effective interventions to minimize bone loss is crucial for comprehensive treatment of patients who undergo bariatric surgery. Specific Aim 1: To determine the efficacy of zoledronic acid in preventing bone loss associated with sleeve gastrectomy (SG). Bone mineral density (BMD) and bone turnover markers will be measured at baseline and 9 months. The primary outcome is change in BMD as measured by Dual-energy x-ray absorptiometry (DXA). Secondary outcomes are change in BMD as measured by Quantitative Computed Tomography (QCT) and change in the serum bone turnover markers, urinary collagen type 1 cross-linked N-telopeptide (CTX; bone formation marker), serum type 1 procollagen N-terminal (P1NP; bone resorption marker), sclerostin, and osteocalcin. Specific Aim 2: To evaluate the feasibility of this trial in those who have undergone SG surgery. The feasibility will be assessed by documenting adverse events and compliance rates of the intervention at each study time point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects planning a sleeve gastrectomy procedure at the University of Nebraska Medical Center (UNMC) Bariatric Center
* Agreement to all study procedures and assessments
* Women must be postmenopausal (FSH blood level > 30 mIU/m), or incapable of child-bearing

Exclusion Criteria:

* Prior bariatric surgery
* < 19 years of age
* Weight ≥ 350lbs
* Liver or renal disease
* Hypercalcemia, hypocalcemia, or hypomagnesemia
* Serum 25-OH vitamin D < 20 ng/mL
* History of bone-modifying disorders
* Use of bone-active medications
* Known sensitivity to bisphosphonates
* Extensive dental work involving extraction or dental implant within the past 2 months or planned in the upcoming 6 months
* Current diagnosis of type 1 diabetes
* Current malignancy
* Autoimmune disease impacting bone (ex: Rheumatoid Arthritis)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Bilek, PT, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Bariatric Center, Nebraska Medicine, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers should contact the study PI for potential access to the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 06/30/2024
Access Criteria: Approval from the PI

REFERENCES:
- [Derived] Flores LE, Mack L, Wichman C, Weaver AA, Kothari V, Bilek LD. Protocol for a pilot randomised controlled trial of zoledronic acid to prevent bone loss following sleeve gastrectomy surgery. BMJ Open. 2021 Dec 9;11(12):e057483. doi: 10.1136/bmjopen-2021-057483. PMID 34887285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Infusion | Non-active Infusion
Started | 3 | 7
Completed | 2 | 7
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Infusion | Non-active Infusion | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Continuous [Median (Full Range); unit: years] | 49.8 [43.9 to 58.7] | 43.1 [35.5 to 66.4] | 44.4 [35.5 to 66.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 7 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 10
Hip BMD [Median (Full Range); unit: g/cm2] | 1.2 [1.1 to 1.4] | 1.2 [1.2 to 1.4] | 1.2 [1.1 to 1.4]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hip Bone Mineral Density (BMD)
Description: Change in hip bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA) - g/cm2
Time Frame: baseline and 10 months post-surgery
Population: Study participants who completed the study
Measure: Median (Full Range); unit: g/cm2
Arm/Group | Active Infusion | Non-active Infusion
Number analyzed (Participants) | 2 | 7
g/cm2 | 0 [-.01 to .01] | -.03 [-.07 to .03]

2. Secondary Outcome: Change in Lumbar Spine Bone Mineral Density (BMD)
Description: Change in lumbar spine bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA)/cm2 of L1-L4 lumbar vertebrae
Time Frame: baseline and 10 months post-surgery
Population: Participants who completed the study
Measure: Median (Full Range); unit: g/cm2
Arm/Group | Active Infusion | Non-active Infusion
Number analyzed (Participants) | 2 | 7
g/cm2 | .06 [.06 to .07] | .06 [-.06 to .09]

3. Secondary Outcome: Change in Trunk Lean Mass
Description: Change in trunk lean mass, measured in kg
Time Frame: baseline and 9 months post-surgery
Population: Participants who completed the study
Measure: Median (Full Range); unit: kg
Arm/Group | Active Infusion | Non-active Infusion
Number analyzed (Participants) | 2 | 7
kg | -2.7 [-3.6 to -1.8] | -3.3 [-4.4 to -1.1]

4. Secondary Outcome: Change in Trunk Fat Mass
Description: Change in Trunk fat mass, measured in kg
Time Frame: baseline and 9 months post-surgery
Population: Participants who completed the study
Measure: Median (Full Range); unit: kg
Arm/Group | Active Infusion | Non-active Infusion
Number analyzed (Participants) | 2 | 7
kg | -1.0 [-5.3 to 3.2] | -5.4 [-8.1 to -1.7]

5. Secondary Outcome: Change in Weight
Description: Change in weight, measured in kgs
Time Frame: baseline and 9 months post-surgery
Population: participants who completed the study
Measure: Median (Full Range); unit: kg
Arm/Group | Active Infusion | Non-active Infusion
Number analyzed (Participants) | 2 | 7
kg | -10.9 [-21.8 to 0.0] | -22.7 [-40.4 to -15.4]

6. Other Pre Specified Outcome: Proportion of Participants Completing 9 Month Study Visit Requirements
Description: Feasibility assessment: proportion of participants completing 9 Month study visit requirements
Time Frame: 9 Months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Tolerance: Total Number of Adverse Events Reported by Participants in the Active and In-active Arms
Description: Comparison of the total number of adverse events reported by participants in the active and in-active arms
Time Frame: 9 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from individual participants during their participation in the study, approximately 10 months.
Arm/Group | Active Infusion | Non-active Infusion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/7
Other Adverse Events (participants affected / at risk) | 0/3 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Infusion (N=3) | Non-active Infusion (N=7)
Surgical Complication (Surgical and medical procedures) | 1 (1) | 0 (0) — One patient had anastomic leak after surgery. Infusion did not occur due to surgical complication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04279392/Prot_SAP_002.pdf
  • Informed Consent Form (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04279392/ICF_003.pdf